CLINICAL TRIAL: NCT02935426
Title: Comparison of Cyanoacrylate Tissue Adhesives to Polytetrafluoroethylene (PTFE) Sutures in the Donor Site of Connective Tissue Grafts- A Randomized Clinical Trial
Brief Title: Comparison of Cyanoacrylate Adhesives to Sutures in the Palate After Connective Tissue Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Chrysi Stavropoulou, Periodontics Resident, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2016:092
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Wound Closure
Keywords: cyanoacrylate; sutures
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyanoacrylate group (Experimental): Wound closure after harvesting of connective tissue graft in the donor site will be achieved with application of cyanoacrylate tissue adhesive
  Interventions: Device: n-butyl cyanoacrylate and 2-octyl cyanoacrylate
- Suture group (Active Comparator): Wound closure after harvesting of connective tissue graft in the donor site will be achieved with polytetrafluoroethylene (PTFE) continuous interlocking sutures
  Interventions: Device: 5-0 Polytetrafluoroethylene (PTFE) suture

INTERVENTIONS:
Device: n-butyl cyanoacrylate and 2-octyl cyanoacrylate — used in cyanoacrylate group
  Other Names: PeriAcryl®90
  Arms: Cyanoacrylate group
Device: 5-0 Polytetrafluoroethylene (PTFE) suture — used in suture group
  Arms: Suture group

SUMMARY:
Cyanoacrylate tissue adhesives have been successfully used for wound closure. The purpose of this clinical trial is to compare cyanoacrylate tissue adhesives to polytetrafluoroethylene (PTFE) sutures in the donor site of connective tissue grafts. Two groups of volunteers will randomly assigned to one of the two study groups. The wound closure at the palatal donor area will be achieved with polytetrafluoroethylene (PTFE) sutures in one group and with high viscosity cyanoacrylate tissue adhesives on the other group. The surgical procedure will be performed by one of three calibrated periodontics residents. Data will be collected at baseline-day of the surgery and in one week post-operatively. The primary outcome is patient's discomfort from the donor site during the first week after the surgery. Secondary outcomes is the time required for suture placement or cyanoacrylate application, patient's pain from donor and recipient site one week post-operatively, painkillers intake, presence or absence of inflammation and modified EHI early-wound healing index.

DETAILED DESCRIPTION:
A prospective, randomized clinical trial will be conducted to determine whether cyanoacrylate tissue adhesives or sutures are better tolerated by patients receiving soft tissue gum grafts.

Periodontal plastic surgery procedures have become an integral part of periodontal treatment by addressing esthetic and functional demands. Several therapeutic modalities such as free gingival graft, pedicle flaps, connective tissue grafts, grafts combining the two lateral modalities and guided tissue regeneration have been used for covering the denuded roots and augmenting the width and thickness of the keratinized gingiva. Among various surgical techniques, subepithelial connective tissue (SECT) grafts remain the most commonly used and most successful root coverage procedures. The esthetic and functional success of SECT graft techniques is highly predictable and reliable and they have given them a common place in the clinical practice. Subepithelial connective tissue graft procedures require harvesting tissue from a donor area, usually the palate. This addition of another surgical site extends the complexity of the procedure and increases patient discomfort.

Single interrupted or continuous interlocking sutures are suggested at the donor site. Suturing is the most common method of wound closure. Other biomaterials such as staples, adhesive tapes, adhesive glues and fibrin sealants have been used generally to hasten the pace of healing. Adhesives interact with different materials, merge and allow them to remain whole. Cyanoacrylates are bio-adhesives that were discovered by Ardis in 1949 and first used for surgery by Coover et al in 1959. When applied to two opposing, wet, living tissue surfaces, they have the ability to cement them in place. Their general chemical formula is CH2=C(CN)-COOR , where R can be substituted for any alkyl group, ranging from methyl to decyl. They polymerize rapidly within seconds in an exothermic reaction following contact with proteinaceous surfaces to form strong and flexible bonds. Methyl cyanoacrylate was the first glue developed, but tissue toxicity precluded its use. The process of causing histologic toxicity is thought to be related to the byproducts of degradation into cyanoacetate and formaldehyde. Further research showed that changing the type of alkyl chains in the compound to one with a longer molecular chain can reduce tissue toxicity. Cyanoacrylates are simple, inexpensive and practical adhesives. Cyanoacrylates have been used for achieving hemostasis at intraoral and extra-oral surgical sites treating ulcers, attaching grafts, managing cerebral spinal fluid leaks, stabilizing the bone fragments during plating, sealing sinus membrane perforations, and achieving peripheral nerve re-anastomosis; as periodontal dressings; and for a number of other dental applications. They are sloughed from the surface of the skin and mucosa 7 to 10 days after adhesive application. Butyl cyanoacrylate is a bacteriostatic, biodegradable, hemostatic cyanoacrylate with a long half-life and good tissue compatibility. It can adhere in moist environments and is available in a formulation appropriate to be used in the oral cavity. It has been proven to be effective in closure of uninfected intraoral incisions on edentulous areas in the mandible, in extractions and periapical surgery.

Few studies are focused on evaluating the wound healing and assessing patient-centered outcomes at the palate donor area after different harvesting techniques To the best of our knowledge, there is no study that compares different methods of wound closure at the donor site.

This prospective clinical trial aims at obtaining information to determine which technique from the patient's standpoint is superior.

The participants will be randomly assigned to one of two groups. The wound closure at the palatal donor area will be achieved with polytetrafluoroethylene (PTFE) sutures in one group and with high viscosity cyanoacrylate tissue adhesives on the other group. The surgical procedure will be performed by one of three calibrated periodontics residents (CS, JB, DR). Patients will be followed for 1 month post-operatively by the same resident to monitor the healing process and obtain patient feedback. Data will be collected at the baseline-day of the surgery, one day post-operatively and at the 1-week follow-up appointment. Randomization will be achieved using a computerized randomization scheme and will be communicated to the surgeon during the surgery by an independent examiner (AC). Participants will be block-randomized for each of the three operators for balance.

Anesthesia will be achieved with greater palatine block anesthesia and local infiltrations, if needed, on the palate with 1.8ml Lidocaine 2% 1:100,000 epinephrine. The single incision harvesting technique is chosen. Following administration for local anesthesia a single incision is made on the anterior hard palatal vault. The length of the incision depends on the size of the graft that is needed.

Once the graft is harvested pressure is applied to the palate until hemostasis is achieved and the graft is maintained in a moist environment.

Using 5-0 PTFE suture, continuous interlocking sutures 4mm apart are placed in the suture group leaving 3-4mm tails. Thin layers of cyanoacrylate are applied and rinsed with saline at least 3 times with interval at least 30s to allow complete polymerization in the cyanoacrylate group until hemostasis is achieved.

The harvested tissue graft is sutured to the donor site. The day of the surgery-a baseline record is obtained (see attached form). A loading dose of Amoxicillin 2g or Clindamycin 600mg, in case of allergy to penicillin, is provided to all participants immediately after the surgery with Ibuprofen 400mg for pain control. Postoperative instructions are also provided. They are also provided with an ice pack for the first 24 hours to minimize swelling from the recipient site. Sufficient amount of Ibuprofen 200mg is provided in a bag for the participants to consume 1-2 tablets po q4-6h PRN. They are instructed to return the bag for recording of the number of painkillers consumed at the 1-week follow-up appointment. A pain visual analogue scale (VAS) questionnaire with no pain on the left site and unbearable pain on the right site is given to the participants to note the level of pain from the palatal site the day after the surgery before the consumption of any painkillers. Participants are encouraged to contact the operator if they have any problem at any time.

Post-operative complications like severe bleeding, infection, abnormal pain, root exposure of the teeth adjacent to the donor site or sloughing, that need to be addressed before the scheduled appointments, will be recorded for 1 month after the surgery.

At the 1-week follow-up appointments the modified early-wound healing index (EHI), the wound length and width, and the presence of normal or abnormal inflammation will be recorded. The number of painkillers consumed the 1st week after the surgery will be counted and recorded. Participants will be asked to report any self-medication for pain. Sutures will be removed in the suture group. A 1-week follow-up VAS questionnaire is given to participants to fill during the 1-week follow-up appointment. The participants are asked to note the level of pain from the donor and recipient site and the level of discomfort (eating, speaking,.) from the donor site during the week after the surgery. Photos will be taken in all appointments.)

ELIGIBILITY:
Inclusion Criteria:

* Patients of the Graduate Periodontics Clinic, College of Dentistry, University of Manitoba that require harvesting of subepithelial connective tissue graft from the palate from October 2016 to December 2017 and have signed the consent form.

Exclusion Criteria:

* Patients with coagulation disorders (Hemophilia a/b, von Willebrand disease, liver disease, anticoagulative therapy), patients on corticosteroids, patients with uncontrolled diabetes mellitus or with any systematic disease that periodontal surgery is contraindicated, and patient with history of contact dermatitis to formaldehyde will be excluded from the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Patient's discomfort from the donor site | During the first week after the surgery
  VAS questionnaire

SECONDARY OUTCOMES:
Operative time | A baseline-during the surgery
  Time required to place sutures or to apply cyanoacrylate tissue adhesives
Pain from the donor site | one day after the surgery
  VAS questionnaire
Pain from donor site | During the first week after the surgery
  VAS questionnaire
Painkillers intake | during the first week after the surgery
  amount of Ibuprofen consumed during the first week after the surgery
modified EHI early-wound healing index | one week post-operatively
  assessment of wound closure and presence of fibrin and/or necrosis
Complications | one week post-operatively
  severe bleeding (more than 20 min), infection (swollen and presence of pus), abnormal pain (maximum consumption of painkillers, self-medication), root exposure, sloughing, other

CONTACTS AND LOCATIONS:
Overall Officials: Chrysi Stavropoulou, DDS, Principal Investigator — University of Manitoba
Locations (1):
- Graduate Periodontics Clinic University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Caffesse RG, Guinard EA. Treatment of localized gingival recessions. Part II. Coronally repositioned flap with a free gingival graft. J Periodontol. 1978 Jul;49(7):357-61. doi: 10.1902/jop.1978.49.7.357. PMID 279663
- [Result] Guinard EA, Caffesse RG. Treatment of localized gingival recessions. Part I. Lateral sliding flap. J Periodontol. 1978 Jul;49(7):351-6. doi: 10.1902/jop.1978.49.7.351. PMID 279662
- [Result] Langer B, Langer L. Subepithelial connective tissue graft technique for root coverage. J Periodontol. 1985 Dec;56(12):715-20. doi: 10.1902/jop.1985.56.12.715. PMID 3866056
- [Result] Cortellini P, Tonetti MS. Clinical performance of a regenerative strategy for intrabony defects: scientific evidence and clinical experience. J Periodontol. 2005 Mar;76(3):341-50. doi: 10.1902/jop.2005.76.3.341. PMID 15857066
- [Result] Pini Prato G, Tinti C, Vincenzi G, Magnani C, Cortellini P, Clauser C. Guided tissue regeneration versus mucogingival surgery in the treatment of human buccal gingival recession. J Periodontol. 1992 Nov;63(11):919-28. doi: 10.1902/jop.1992.63.11.919. PMID 1453307
- [Result] Chambrone L, Tatakis DN. Periodontal soft tissue root coverage procedures: a systematic review from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S8-51. doi: 10.1902/jop.2015.130674. PMID 25644302
- [Result] Pandit N, Khasa M, Gugnani S, Malik R, Bali D. Comparison of two techniques of harvesting connective tissue and its effects on healing pattern at palate and recession coverage at recipient site. Contemp Clin Dent. 2016 Jan-Mar;7(1):3-10. doi: 10.4103/0976-237X.177099. PMID 27041892
- [Result] Fickl S, Fischer KR, Jockel-Schneider Y, Stappert CF, Schlagenhauf U, Kebschull M. Early wound healing and patient morbidity after single-incision vs. trap-door graft harvesting from the palate--a clinical study. Clin Oral Investig. 2014 Dec;18(9):2213-9. doi: 10.1007/s00784-014-1204-7. Epub 2014 Feb 23. PMID 24562700
- [Result] Vastani A, Maria A. Healing of intraoral wounds closed using silk sutures and isoamyl 2-cyanoacrylate glue: a comparative clinical and histologic study. J Oral Maxillofac Surg. 2013 Feb;71(2):241-8. doi: 10.1016/j.joms.2012.08.032. Epub 2012 Oct 22. PMID 23089654
- [Result] Gumus P, Buduneli E. Graft stabilization with cyanoacrylate decreases shrinkage of free gingival grafts. Aust Dent J. 2014 Mar;59(1):57-64. doi: 10.1111/adj.12149. Epub 2014 Feb 4. PMID 24494804
- [Result] Costa HJ, Pereira CS, Costa MP, Fabri FS, Lancellotti CL, Dolci JE. Experimental comparative study in rabbits of three different ways of cartilage graft fixation: suture, gelatin-resorcin-formaldehyde and butyl-2-cyanoacrylate. Acta Otolaryngol. 2007 Sep;127(9):947-51. doi: 10.1080/00016480601089689. PMID 17712674
- [Result] Yoo J, Chandarana S, Cosby R. Clinical application of tissue adhesives in soft-tissue surgery of the head and neck. Curr Opin Otolaryngol Head Neck Surg. 2008 Aug;16(4):312-7. doi: 10.1097/MOO.0b013e3283018209. PMID 18626248
- [Result] Leggat PA, Kedjarune U, Smith DR. Toxicity of cyanoacrylate adhesives and their occupational impacts for dental staff. Ind Health. 2004 Apr;42(2):207-11. doi: 10.2486/indhealth.42.207. PMID 15128170
- [Result] Toriumi DM, Raslan WF, Friedman M, Tardy ME. Histotoxicity of cyanoacrylate tissue adhesives. A comparative study. Arch Otolaryngol Head Neck Surg. 1990 May;116(5):546-50. doi: 10.1001/archotol.1990.01870050046004. PMID 2183824
- [Result] Forrest JO. The use of cyanoacrylates in periodontal surgery. J Periodontol. 1974 Apr;45(4):225-9. doi: 10.1902/jop.1974.45.4.225. No abstract available. PMID 4594350
- [Result] Herod EL. Cyanoacrylates in dentistry: a review of the literature. J Can Dent Assoc. 1990 Apr;56(4):331-4. PMID 2196101
- [Result] Habib A, Mehanna A, Medra A. Cyanoacrylate: a handy tissue glue in maxillofacial surgery: our experience in alexandria, egypt. J Maxillofac Oral Surg. 2013 Sep;12(3):243-7. doi: 10.1007/s12663-012-0433-z. Epub 2012 Sep 15. PMID 24431849
- [Result] Ghoreishian M, Gheisari R, Fayazi M. Tissue adhesive and suturing for closure of the surgical wound after removal of impacted mandibular third molars: a comparative study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Jul;108(1):e14-6. doi: 10.1016/j.tripleo.2009.03.001. Epub 2009 May 22. PMID 19464207
- [Result] Sachs HA, Farnoush A, Checchi L, Joseph CE. Current status of periodontal dressings. J Periodontol. 1984 Dec;55(12):689-96. doi: 10.1902/jop.1984.55.12.689. PMID 6394736
- [Result] Kulkarni S, Dodwad V, Chava V. Healing of periodontal flaps when closed with silk sutures and N-butyl cyanoacrylate: a clinical and histological study. Indian J Dent Res. 2007 Apr-Jun;18(2):72-7. doi: 10.4103/0970-9290.32424. PMID 17502712
- [Result] Kondoh S, Matsuo K, Yuzuriha S, Kikuchi N, Ban R. Dressing for alveolopalatal wounds after alveolar bone grafting. Ann Plast Surg. 2003 Sep;51(3):290-3. doi: 10.1097/01.SAP.0000063757.61972.54. PMID 12966242
- [Result] Perez M, Fernandez I, Marquez D, Bretana RM. Use of N-butyl-2-cyanoacrylate in oral surgery: biological and clinical evaluation. Artif Organs. 2000 Mar;24(3):241-3. doi: 10.1046/j.1525-1594.2000.06519.x. PMID 10759649
- [Result] Al-Belasy FA, Amer MZ. Hemostatic effect of n-butyl-2-cyanoacrylate (histoacryl) glue in warfarin-treated patients undergoing oral surgery. J Oral Maxillofac Surg. 2003 Dec;61(12):1405-9. doi: 10.1016/j.joms.2002.12.001. PMID 14663804
- [Result] Lorenzana ER, Allen EP. The single-incision palatal harvest technique: a strategy for esthetics and patient comfort. Int J Periodontics Restorative Dent. 2000 Jun;20(3):297-305. PMID 11203571
- [Result] Wachtel H, Schenk G, Bohm S, Weng D, Zuhr O, Hurzeler MB. Microsurgical access flap and enamel matrix derivative for the treatment of periodontal intrabony defects: a controlled clinical study. J Clin Periodontol. 2003 Jun;30(6):496-504. doi: 10.1034/j.1600-051x.2003.00013.x. PMID 12795787
- [Result] Ronis ML, Harwick JD, Fung R, Dellavecchia M. Review of cyanoacrylate tissue glues with emphasis on their otorhinolaryngological applications. Laryngoscope. 1984 Feb;94(2 Pt 1):210-3. doi: 10.1288/00005537-198402000-00012. PMID 6694493